CLINICAL TRIAL: NCT05715541
Title: Inr Tracking With Face-To-Face And Phone App: A Randomized Controlled Trial
Brief Title: Inr Tracking Coumadin Use With Phone App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed Onur Hanedan (Other)
Responsible Party: Principal Investigator, Muhammet Onur HANEDAN, MD, Associate Professor, Muhammed Onur Hanedan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20/01/2021-2021/15-01
Record Dates: First submitted 2023-01-18; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Warfarin; Mobile Applications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparison of INR Control and Drug Compliance Values by Groups (Other): Follow-up of the patients in the control group continued in the outpatient clinic.
  This application includes an interface where patients can enter drug treatment information such as INR values, disease diagnosis, how many times a day and how many mg they take, and a chat box section where they can communicate with their physicians, including emergencies. The doctor reviewed the patient's INR findings once they were relayed by the patient, then told them to adjust the patient's warfarin dosage and schedule the next INR check. The application sent notifications to the patients every day about when and how many mg of the drug they would take
  Interventions: Other: mobile applications with the name "Set My INR"

INTERVENTIONS:
Other: mobile applications with the name "Set My INR" — The relevant software company assisted in developing the phone application. The language of the application created with the name "Set My INR" is Turkish. The application provided an opportunity for patients to share and communicate with their physician after having the INR value measured in a health institution near their place of residence before coming to the hospital

SUMMARY:
This study aims to compare the INR values of the patients followed by face-to-face and telephone applications.

DETAILED DESCRIPTION:
Warfarin has a narrow therapeutic window. Maintaining the patient's international normalized ratio (INR) within the predefined therapeutic range is one of the main challenges of warfarin treatment. This study was designed as a randomized controlled experiment. Twelve patients living in a distant place were assigned to the experimental group, and 12 patients living nearby and followed in the outpatient clinic were assigned to the control group. A Patient Information Form and the Adherence to Refills and Medications Scale were used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old, using a smartphone, not having a psychiatric illness or treatment, and agreeing to participate

Exclusion Criteria:

* requiring medical examination, not using a smartphone, having a psychiatric illness or treatment, and not agreeing to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the Knowledge Levels of the Groups on the Use of Coumadin | It ranges from 6 months to 1 year
  To measure the knowledge level with "Patient Information Form" of patients using coumadin about the medication.
Comparison of INR Control and Drug Compliance Values by Groups | It ranges from 6 months to 1 year
  Measuring medication compliance with "The Adherence to Refills and Medications Scale" of patients using coumadin.
  To compare the INR values of the patients using the phone application and followed face to face.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Onur HANEDAN, Principal Investigator — MD, Associate Professor1
Locations (1):
- Ahi Evren Göğüs Kalp ve Damar Cerrahisi Eğitim ve Araştırma Hastanesi, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.